CLINICAL TRIAL: NCT04593524
Title: The Role of Vitamin D, A, and Beta Carotene in Tuberculosis Patients With Vitamin D Receptor Gene Polymorphism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Sumatera Utara (Other)
Responsible Party: Principal Investigator, DINA KEUMALA SARI, Principal Investigator, Universitas Sumatera Utara
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: USU 2
Record Dates: First submitted 2020-09-29; First posted 2020-10-20 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Tuberculosis
Keywords: 25(OH)D serum; calcium; counseling; FokI; retinol; TaqI
MeSH Terms: conditions — Tuberculosis | interventions — Vitamin D; Dietary Supplements; Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Active Comparator): 24 participants, which are treatment group (I) which receives nutritional counseling, vitamin D 1000 IU, vitamin A 6000 IU
  Interventions: Dietary Supplement: vitamin D 1000 IU and A 6000 IU supplementation and nutritional counseling
- Counseling Group (Active Comparator): 24 participants which only receives nutritional counseling for 28 days
  Interventions: Other: nutritional Counseling

INTERVENTIONS:
Dietary Supplement: vitamin D 1000 IU and A 6000 IU supplementation and nutritional counseling — 24 participants, which are treatment group (I) which receives nutritional counseling, vitamin D 1000 IU, vitamin A 6000 IU
  Arms: Treatment Group
Other: nutritional Counseling — control group (C) which only receives nutritional counseling for 28 days
  Arms: Counseling Group

SUMMARY:
Recent studies showed that vitamin D and A has an effect in improving sputum conversion in tuberculosis. This study aims to find out the effect of vitamin D 1000 IU and A 6000 IU supplementation on Tuberculosis patients with vitamin D receptor gene polymorphism, who live in North Sumatera, Indonesia. This study is a randomized control clinical trial, with 48 tuberculosis patients with vitamin D receptor gene polymorphism which are TaqI and FokI participating, divided into two groups, each with 24 participants, which are treatment group (I) which receives nutritional counseling, vitamin D 1000 IU, vitamin A 6000 IU, and control group (C) which only receives nutritional counseling for 28 days. Patients who participated was found to be heterozygous with TaqI (T>C) or FokI (C>T) genotype variants.

DETAILED DESCRIPTION:
Recent studies showed that vitamin D and A has an effect in improving sputum conversion in tuberculosis. This study aims to find out the effect of vitamin D 1000 IU and A 6000 IU supplementation on Tuberculosis patients with vitamin D receptor gene polymorphism, who live in North Sumatera, Indonesia. This study is a randomized control clinical trial, with 48 tuberculosis patients with vitamin D receptor gene polymorphism which are TaqI and FokI participating, divided into two groups, each with 24 participants, which are treatment group (I) which receives nutritional counseling, vitamin D 1000 IU, vitamin A 6000 IU, and control group (C) which only receives nutritional counseling for 28 days. Patients who participated was found to be heterozygous with TaqI (T>C) or FokI (C>T) genotype variants. The result of this study showed that at the start, serum 25(OH)D levels in group I were lower compared to group C (19.746.59 ng/mL vs 25.21±7.57 ng/mL). Group I showed significant correlation between vitamin D level categories with sputum conversion (mean: standard deviation= 2.25±0.68 weeks). Supplementation of vitamin D 1000 IU provides an accelerated sputum conversion in tuberculosis patients with vitamin D receptor gene polymorphism.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria are males or females, which have new case lung tuberculosis infection with acid fast bacilli (AFB) result (+), aged 18-60 years, heterozygote genotype test on one of the genes TaqI and FokI, willing to participate in the study and complete the informed consent.

Exclusion Criteria:

* The exclusion criteria are pregnant, found to have comorbidities such as diabetes mellitus or Human Immunodeficiency Virus (+), and Tuberculosis on category II.

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Mrs / Miss
Enrollment: 48 (Actual)
Dates: Start 2019-05-14 (Actual); Primary Completion 2019-08-15 (Actual); Study Completion 2019-09-22 (Actual)

PRIMARY OUTCOMES:
vitamin D | up to 4 weeks
  25(OH)D serum level
vitamin A | up to 4 weeks
  vitamin A serum level
beta carotene | up to 4 weeks
  beta carotene

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Universitas Sumatera Utara, Medan, North Sumatra, Indonesia

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-05-09): https://cdn.clinicaltrials.gov/large-docs/24/NCT04593524/Prot_SAP_000.pdf
  • Informed Consent Form (2020-05-09): https://cdn.clinicaltrials.gov/large-docs/24/NCT04593524/ICF_001.pdf